CLINICAL TRIAL: NCT00109720
Title: Evaluation of Diabetes Self-Management Consultant Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Detroit Department of Health (Other)
Responsible Party: Robert M Anderson EdD Professor, University of Michigan Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 62323 (completed)
Record Dates: First submitted 2005-05-02; First posted 2005-05-03 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Self Management; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients in the experimental group received the services of a Diabetes Self-Management Consultant (DSC)
  Interventions: Behavioral: Diabetes Self-Management Consultant
- 2 (Active Comparator): This Arm was a Enhanced Usual Care Control group who continued with their usual care but also they and their physicians received the results of all metabolic assessments obtained during the study.
  Interventions: Behavioral: Enhanced Usual Care Control Group

INTERVENTIONS:
Behavioral: Diabetes Self-Management Consultant — services of a Diabetes Self-Management Consultant
  Arms: 1
Behavioral: Enhanced Usual Care Control Group — Usual care plus results of metabolic assessments obtained during the study
  Arms: 2

SUMMARY:
The purpose of this study is to find out if Self-Management Consultant (SMC) intervention will be more effective than usual care in improving blood glucose control and diabetes-related quality of life for adults with type 2 diabetes.

DETAILED DESCRIPTION:
This study is designed to compare the effectiveness of a diabetes Self-Management Consultant (SMC) intervention for adults with type 2 diabetes with unsatisfactory glucose control (i.e., HbA1c ≥ 8%--the value chosen as "high risk" by the Diabetes Quality Improvement Project which is an initiative of the Health Care Financing Administration, the American Diabetes Association, and the Foundation for Accountability) to a control group selected using the same criteria. The SMC intervention will be implemented and evaluated in two different health care systems serving two distinct populations of patients with diabetes. After signing the Informed Consent document, subjects will be randomized to the SMC intervention or a control group. All subjects in the study will complete a baseline assessment of their diabetes care and health status.

Subjects randomized to the SMC intervention will have an individual meeting with the SMC to review and refine a self-management plan based on the subject's priorities and goals. These subjects will receive individual follow-up and support during the year, through monthly phone calls and an annual meeting with the SMC and their primary care physician. Subjects randomized to the control group will receive usual care following their baseline and their 12-, 24-, and 36-month assessments. Unlike most nurse-manager studies, the SMC's interactions with patient care will use a theory-based behavioral approach with which we have extensive experience. The study is designed to evaluate the effectiveness of the SMC intervention compared to usual care.

All records will be handled confidentially. Lab results and personal data will be linked by a research specific identifier code.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age 21 diagnosed with type 2 diabetes for at least one year.

Exclusion Criteria:

* Patients under psychiatric care
* Currently pregnant
* Those who have not been diagnosed with type 2 diabetes

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2002-08; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Blood glucose level | two years

SECONDARY OUTCOMES:
Diabetes Related Quality of life | two years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Anderson, Ed. D., Principal Investigator — Department of Medical Education, University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Department of Family Medicine Clinics, Ann Arbor, Michigan
  - Detroit Health Department, Detroit, Michigan

REFERENCES:
- [Background] Heisler M, Vijan S, Anderson RM, Ubel PA, Bernstein SJ, Hofer TP. When do patients and their physicians agree on diabetes treatment goals and strategies, and what difference does it make? J Gen Intern Med. 2003 Nov;18(11):893-902. doi: 10.1046/j.1525-1497.2003.21132.x. PMID 14687274
- [Background] Funnell MM, Anderson RM. Changing office practice and health care systems to facilitate diabetes self-management. Curr Diab Rep. 2003 Apr;3(2):127-33. doi: 10.1007/s11892-003-0036-7. PMID 12728638
- [Background] Funnell MM, Anderson RM. Patient empowerment: a look back, a look ahead. Diabetes Educ. 2003 May-Jun;29(3):454-8, 460, 462 passim. doi: 10.1177/014572170302900310. No abstract available. PMID 12854337
- [Background] Anderson RM, Fitzgerald JT, Gruppen LD, Funnell MM, Oh MS. The Diabetes Empowerment Scale-Short Form (DES-SF). Diabetes Care. 2003 May;26(5):1641-2. doi: 10.2337/diacare.26.5.1641-a. No abstract available. PMID 12716841
- [Background] Funnell MM, Anderson RM. Working toward the next generation of diabetes self-management education. Am J Prev Med. 2002 May;22(4 Suppl):3-5. doi: 10.1016/s0749-3797(02)00431-2. No abstract available. PMID 11985929
- [Background] Anderson RM, Funnell MM. Compliance and adherence are dysfunctional concepts in diabetes care. Diabetes Educ. 2000 Jul-Aug;26(4):597-604. doi: 10.1177/014572170002600405. PMID 11140071